CLINICAL TRIAL: NCT03643718
Title: Web-based International Register of Emergency Surgery and Trauma
Acronym: WIRES-T
Status: Recruiting | Type: Observational
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: World Society of Emergency Surgery (Other); University of Pisa (Other)
Responsible Party: Principal Investigator, Federico Coccolini, MD, Attending Surgeon, University of Pisa
Other Study IDs: FC-001-2018
Record Dates: First submitted 2018-05-14; First posted 2018-08-23 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Acute Appendicitis; Acute Cholecystitis; Acute Diverticulitis; Post-operative Complications; Acute Pancreatitis; Perforated Gastro-duodenal Ulcers; Adhesive Small Bowell Occlusion; Colonic Neoplastic Emergencies; Gynecological Emergencies; Vascular Emergencies; Intestinal Ischemia; Abdominal Wall Hernia; Foreign Bodies; Caustic Ingestion; Trauma
MeSH Terms: conditions — Appendicitis; Cholecystitis, Acute; Pancreatitis; Hernia, Abdominal; Foreign Bodies; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Emergency General Surgery — Emergency General Surgery and Trauma operative/non operative management
  Other Names: Trauma

SUMMARY:
The WIRES-T project (Web-based International Registry of Emergency General Surgery and Trauma) has been set up to allow to all the EGS (Emergency General Surgery) and Trauma surgeons to register their activity and to obtain a worldwide register of traumatic and non traumatic surgical emergencies. This will give the opportunity to evaluate results on a macro-data basis and to give index allowing stratifying, evaluating and improving the outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by an acute surgical disease
* Patients with indication to be referred to the emergency surgeon attention
* Patients to be operated or to be treated with non-operative approach without surgical intervention

Exclusion Criteria:

* Patients not affected by an acute surgical disease
* Patients without indication to be referred to the emergency surgeon attention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients affected by an acute surgical disease and/or who may require to be undergone to the emergency surgeon attention to be managed either with an operative or a non-operative approach.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Rate of patients treated with surgery | Until hospital discharge, approximately 2 weeks
  Evaluate the rate of operative treatment for each different disease according to the different enviroment; for each intervention the surgical approach (laparotomic, mini-invasive, laparoscopic) will be evaluated.
Rate of patients treated with conservative treatment | Until hospital discharge, approximately 2 weeks
  Evaluate the conservative treatment rate for each different disease according to patient's characteristics and the enviroinment.

SECONDARY OUTCOMES:
Mortality | Until hospital discharge, approximately 2 weeks
  To evaluate the differences in mortality rate linked to the different managements, techniques, environments and patient variables.
Morbidity | Until hospital discharge, approximately 2 weeks
  To evaluate the differences in morbidity rate linked to the different managements, techniques, environments and patient variables.

CONTACTS AND LOCATIONS:
Locations (1):
- General, Emergency and Trauma surgery, University Hospital of Pisa, Pisa, Italy

REFERENCES:
- [Derived] Coccolini F, Mazzoni A, Cremonini C, Cobuccio L, Pucciarelli M, Vetere G, Borelli B, Strambi S, Musetti S, Miccoli M, Cremolini C; WIRES-T Study Group; Tartaglia D, Chiarugi M. Colorectal neoplastic emergencies in immunocompromised patients: preliminary result from the Web-based International Register of Emergency Surgery and Trauma (WIRES-T trial). Updates Surg. 2023 Sep;75(6):1579-1587. doi: 10.1007/s13304-023-01521-8. Epub 2023 May 9. PMID 37160552